CLINICAL TRIAL: NCT04964492
Title: Assessment of the Hemodynamic Effect of Hydroxocabalamin in Refractory Vasodilatory Shock
Acronym: VASOKIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0124
Record Dates: First submitted 2021-07-13; First posted 2021-07-16 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Vasoplegia; Hemodynamics; Intensive Care Unit; Shock
Keywords: vasoplegia; hydroxocobalamin; hemodynamics; intensive care unit; shock
MeSH Terms: conditions — Vasoplegia; Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- responders to treatment: A patient will be defined as a responder to hydroxocobolamin infusion if there is an increase of more than 20% in Average blood pressure, relative to the pre-treatment value, for at least 15 minutes within one hour of treatment administration.
- non-responders to treatment: A patient will be defined as a non-responder to hydroxocobolamin infusion if there is not an increase of more than 20% in Average blood pressure, relative to the pre-treatment value, for at least 15 minutes within one hour of treatment administration.

SUMMARY:
Through clinical cases or retrospective work with small sample size, some authors have observed an improvement in hemodynamic parameters, with a reduction or even withdrawal of norepinephrine after administration of a single dose of hydroxocobolamin (HCB) in refractory vasoplegic shock (cardiac surgery, liver transplantation and septic shock).

HCB produces beneficial alterations in NO metabolism and may be suitable in vasoplegic syndrome. In addition, HCB seems to be involved in the elimination of hydrogen sulfide which also has an endogenous vasodilator function in the vascular endothelium. By these different actions it would cause vasoconstriction in vascular smooth muscle cells. Previous reports demonstrate that HCB was useful for refractory vasoplegic syndrome.

The investigators will conduct a retrospective data collection of patients who was given intravenous HCB for refractory vasoplegic shock since January 2019.

DETAILED DESCRIPTION:
Vasoplegic shock is defined by arterial hypotension, a high cardiac output with a normal or high cardiac index, collapsed systemic vascular resistance (SVR) and high dose of norepinephrine in the absence of hypovolaemia. The drop in secondary organ perfusion pressure ultimately leads to multiple organ failure and death.

Through clinical cases or retrospective work with small sample size, some authors have observed an improvement in hemodynamic parameters, with a reduction or even withdrawal of norepinephrine after administration of a single dose of hydroxocobolamin (HCB) in refractory vasoplegic shock (cardiac surgery, liver transplantation and septic shock).

HCB produces beneficial alterations in NO metabolism and may be suitable in vasoplegic syndrome. In addition, HCB seems to be involved in the elimination of hydrogen sulfide which also has an endogenous vasodilator function in the vascular endothelium. By these different actions it would cause vasoconstriction in vascular smooth muscle cells. Previous reports demonstrate that HCB was useful for refractory vasoplegic syndrome.

The investigators will conduct a retrospective data collection of patients who was given intravenous HCB for refractory vasoplegic shock since January 2019.

ELIGIBILITY:
Inclusion Criteria:

* All SVR patients over 18 years of age who had received a dose of HCB since January 1 2019 will be included.

Exclusion Criteria:

* Patients who received treatment for another indication were not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All SVR (systemic vascular resistance) patients over 18 years of age who had received a dose of HCB since January 1 2019 will be included. Patients who received treatment for another indication were not included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients responding to treatment with HCB | 1 hour
  A patient will be defined as a responder to hydroxocobalamin infusion if there is an increase of more than 20% in average blood pressure, relative to the pre-treatment value, for at least 15 minutes within one hour of treatment administration.

SECONDARY OUTCOMES:
The change in average blood pressure over time in responder patients | one hour
  Blood pressure is measured in units of millimeters of mercury (mmHg).
The change in average blood pressure over time in non-responder patients | one hour
  Blood pressure is measured in units of millimeters of mercury (mmHg).
The change in doses of NAd (mg/h) in responder patients | one hour
The change in doses of NAd (mg/h) in non-responder patients | one hour

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No